CLINICAL TRIAL: NCT07170709
Title: Effect of Mechanical Load Magnitude on Reflex Latency Induced by Whole-Body Vibration: A Latency-Based Evaluation of Bone Myoregulation Reflex and Tonic Vibration Reflex
Brief Title: WBV Reflex Latency and Mechanical Load
Acronym: WBV-BMR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selim Sezikli (Other Government)
Responsible Party: Sponsor-Investigator, Selim Sezikli, Principal Investigator / Physical Medicine & Rehabilitation Specialist, Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Organization: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: WBV-BMR-2025-01; 2017.124.IRB2.038 (Other: Koç University IRB)
Record Dates: First submitted 2025-08-29; First posted 2025-09-12 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-08

CONDITIONS: Whole-body Vibration; Healthy Volunteers (HV); Muscle Contraction; Postural Balance; Electromyography
Keywords: Whole-Body Vibration; Tonic Vibration Reflex; Bone Myoregulation Reflex; Reflex Latency; Postural Reflexes; Surface Electromyography; Mechanical Loading; Healthy Volunteers; Neuromuscular Physiology

STUDY DESIGN:
Intervention Model Description: All participants receive the same sequence of whole-body vibration under different loading conditions. There is no randomization or control group. This is a single-arm, within-subject experimental design evaluating reflex latency under multiple biomechanical scenarios.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Whole-Body Vibration in Healthy Volunteers (Experimental): Participants will receive whole-body vibration (WBV) under mechanical loading conditions. Surface EMG recordings from the soleus muscle will be used to evaluate reflex latency at vibration frequencies of 30, 32, 34, and 36 Hz. All interventions will be applied in a single-session experimental design in healthy adult volunteers.
  Interventions: Device: Whole-Body Vibration

INTERVENTIONS:
Device: Whole-Body Vibration — Participants will receive whole-body vibration (WBV) at 30-36 Hz under different mechanical loading conditions (e.g., standing on one foot, both feet,). Vibration-induced reflex responses will be recorded from the soleus muscle using surface electromyography. The intervention is designed to evaluate latency differences between tonic vibration reflex (TVR) and bone myoregulation reflex (BMR) under controlled biomechanical scenarios.
  Other Names: WBV; Reflex Latency Vibration Protocol

SUMMARY:
This study aims to investigate how the magnitude of mechanical loading affects reflex latency patterns induced by whole-body vibration (WBV). WBV can trigger two types of reflexes: the tonic vibration reflex (TVR) and the bone myoregulation reflex (BMR), which may be influenced by load-bearing condition. The study will include healthy adult volunteers aged 20-50 years. Reflex responses will be recorded from the soleus muscle using surface EMG during both WBV. Different conditions of mechanical loading (i.e., standing on one foot, both feet) and vibration frequencies (30-36 Hz) will be tested. The main outcome will be the latency of the reflex responses, which will help distinguish between TVR and BMR activation. The goal is to better understand how mechanical load modifies reflex response timing and to characterize the underlying afferent pathways. This knowledge may contribute to optimizing vibration-based rehabilitation strategies.

DETAILED DESCRIPTION:
This study investigates how the magnitude of mechanical loading alters reflex latency patterns during whole-body vibration (WBV), focusing specifically on the tonic vibration reflex (TVR) and the bone myoregulation reflex (BMR). Experimental data suggest that WBV may activate different reflex mechanisms depending on the level of postural loading, frequency, and amplitude of the vibration. Previous studies have shown that low-amplitude WBV tends to activate TVR under voluntary contraction, while higher mechanical loads and neutral standing posture are more likely to induce BMR.

Surface electromyography (sEMG) recordings will be obtained from the soleus muscle during vibration stimuli applied at different frequencies (30, 32, 34, and 36 Hz). Recordings will be taken under multiple loading conditions: standing on both feet, standing on one foot. Reflex latency will be calculated using cumulative averaging techniques, and data will be analyzed offline using Spike2 software.

Findings from this study may contribute to a deeper understanding of reflex integration during vibratory stimulation and inform future neurorehabilitation protocols that utilize WBV as a therapeutic modality.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 40 years
* Healthy adult volunteers with no known neurological or musculoskeletal disorders
* Able to provide informed consent
* Willing to comply with the procedures of the study, including EMG and vibration exposure

Exclusion Criteria:

* History of any neurological condition (e.g., peripheral neuropathy, spinal cord injury, stroke)
* Musculoskeletal injury or surgery involving the lower extremities
* Use of medications affecting neuromuscular function
* Pregnancy
* Presence of implanted electronic devices (e.g., pacemaker)
* Known intolerance to vibration exposure

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2025-09-02 (Actual); Primary Completion 2025-09-20 (Actual); Study Completion 2025-09-24 (Actual)

PRIMARY OUTCOMES:
Reflex latency (milliseconds) in the soleus muscle during vibration stimulation | Day 1 (single-session, during each experimental condition)
  Reflex latency will be calculated based on surface EMG recordings from the soleus muscle during whole-body vibration at frequencies of 30-36 Hz. Latency will be analyzed using cumulative averaging techniques and expressed in milliseconds.

SECONDARY OUTCOMES:
EMG amplitude of reflex response in the soleus muscle during vibration stimulation | Day 1 (single-session, during each experimental condition)
  The magnitude of EMG response during whole-body vibration will be recorded from the soleus muscle. Reflex amplitude differences will be analyzed across various postural loading conditions to evaluate suppression or facilitation effects.
Reflex type classification (TVR vs BMR) based on latency and mechanical load | Day 1 (single-session, during each experimental condition)
  Reflex responses will be categorized as tonic vibration reflex (TVR) or bone myoregulation reflex (BMR) based on latency values and mechanical loading condition. Classification will be supported by comparisons of reflex latency and EMG suppression patterns across experimental conditions.
Reflex latency variability under different mechanical loading conditions | Day 1 (single-session, during each experimental condition)
  Variability in reflex latency will be assessed across different postural load conditions (e.g., single-leg, double-leg, prone) to determine how load magnitude influences the consistency of reflex timing. Standard deviation and coefficient of variation will be calculated for each condition.
Effect of vibration frequency on reflex latency and amplitude | Day 1 (single-session, during each experimental condition)
  Reflex latency and EMG amplitude will be compared across vibration frequencies (30, 32, 34, and 36 Hz) to investigate frequency-dependent modulation of neuromuscular responses in the soleus muscle.

CONTACTS AND LOCATIONS:
Overall Officials: Selim Sezikli, MD, Principal Investigator — Istanbul Physical Medicine and Rehabilitation Training and Research Hospital
Locations (1):
- Istanbul Physical Medicine and Rehabilitation Training and Research Hospital, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Following publication of the main study results, de-identified individual participant data (IPD) and relevant supporting documents will be made available to qualified researchers upon submission of a valid research proposal. Data will be provided exclusively for research purposes and under a formal data sharing agreement.
Supporting Information: Study Protocol
Time Frame: Data will be available beginning 6 months after the primary publication and will remain accessible for 5 years. Access will be granted on a case-by-case basis following review of a research proposal and execution of a formal data-sharing agreement.
Access Criteria: Access will be limited to qualified researchers who submit a request for a research project that has received prior ethical approval and who agree to comply with the study's confidentiality principles. Data access will be granted through a formal data-sharing agreement executed between the requesting researcher and the study sponsor or relevant institution. The agreement will specify the intended purpose of data use, the duration of access, and the confidentiality obligations. Shared data will consist of de-identified individual participant data (IPD), with all potentially identifying information removed. Supporting documents such as the study protocol, statistical analysis plan, and analytic code will also be provided to promote research transparency.
URL: https://istanbulftr.saglik.gov.tr

REFERENCES:
- [Background] Karacan I, Turker KS. Exploring neuronal mechanisms of osteosarcopenia in older adults. J Physiol. 2026 Jan;604(2):672-688. doi: 10.1113/JP285666. Epub 2024 Aug 9. PMID 39119811
- [Background] Karacan I, Cidem M, Yilmaz G, Sebik O, Cakar HI, Turker KS. Tendon reflex is suppressed during whole-body vibration. J Electromyogr Kinesiol. 2016 Oct;30:191-5. doi: 10.1016/j.jelekin.2016.07.008. Epub 2016 Jul 25. PMID 27485766
- [Background] Karacan I, Cidem M, Cidem M, Turker KS. Whole-body vibration induces distinct reflex patterns in human soleus muscle. J Electromyogr Kinesiol. 2017 Jun;34:93-101. doi: 10.1016/j.jelekin.2017.04.007. Epub 2017 Apr 24. PMID 28457998